CLINICAL TRIAL: NCT00316628
Title: A Phase II, Open Label, Uncontrolled, Multi Center Study to Evaluate Safety and Immunogenicity of a Surface Antigen, Inactivated, (Adjuvanted With MF59C.1) Influenza Vaccine, Formulation 2005-2006, When Administered to Elderly Subjects.
Brief Title: Safety and Immunogenicity of an Adjuvanted Influenza Vaccine in Subjects Aged 65 Years and Over.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V70P3S; Eudract number: 2005-000621-38
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2006-09-14 (Estimated); Status verified 2006-09

CONDITIONS: Influenza
Keywords: influenza; elderly; vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

INTERVENTIONS:
Biological: influenza vaccine

SUMMARY:
The purpose of this study is to evaluate safety and immunogenicity of a single intramuscular (IM) injection of an adjuvanted influenza vaccine in elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older and in good health

Exclusion Criteria:

* Any serious disease such as: cancer, autoimmune disease, advanced arteriosclerotic disease or complicated diabetes mellitus, chronic obstructive pulmonary disease (COPD) that requires oxygen therapy, acute or progressive hepatic disease, acute or progressive renal disease, congestive heart failure.
* any acute disease or infections requiring systemic antibiotic or antiviral therapy
* hypersensitivity to eggs, chicken protein, chicken feathers, influenza viral protein, neomycin or polymyxin or any other component of the vaccine
* history of neurological symptoms or signs, or anaphylactic shock following administration of any vaccine
* known or suspected (or high risk of developing) impairment/alteration of immune function within the past 7 days

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50
Dates: Start 2005-06

PRIMARY OUTCOMES:
CHMP criteria for evaluation of flu vaccines e.g Seroprotection, GMR's and Seroconversion rate at day 21 following vaccination.

SECONDARY OUTCOMES:
Number and percentage of subjects with at least one local reaction between Day 0 and Day 3 after vaccine injection.
Number and percentage of subjects with at least one systemic reaction between Day 0 and Day 3 after vaccine injection.
Number and percentage of subjects with at least one adverse event between Day 0 and the study termination visit (Day 21, window: 20-24).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines - Drug Information Services, Study Director — Novartis
Locations (2):
- Italy (2):
  - G. D'Annunzio University, Chieti
  - Office of Hygiene and Public Health, ASL Lanciano, Lanciano